CLINICAL TRIAL: NCT03998072
Title: Does Five Session CAT (Cognitive Analytic Therapy) Consultancy Lead to Improve Outcomes for Patients and Care Coordinators?
Brief Title: Does Five Session CAT Consultancy Lead to Improved Outcomes?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amrit Sinha (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Amrit Sinha, Research Support Officer, University of Sheffield
Organization: University of Sheffield (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 160787
Record Dates: First submitted 2019-05-28; First posted 2019-06-25 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Psychological Intervention; Treatment as Usual
Keywords: psychology; cognitive analytic therapy

STUDY DESIGN:
Intervention Model Description: The study will utilise two conditions - intervention and waiting list. Participants on the waiting list will then proceed to the intervention condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Five session cognitive analytic therapy (CAT) consultancy
- Treatment as usual (waiting list control) (No Intervention)

INTERVENTIONS:
Other: Five session cognitive analytic therapy (CAT) consultancy — Five session consultancy with patients and care coordinators using cognitive analytic therapy
  Arms: Intervention

SUMMARY:
Five session CAT (Cognitive Analytic Therapy) consultancy was developed for patients whom services 'struggle to help', such as those with diagnoses of personality disorder. Five session CAT consultancy works with both patients and care coordinators, utilising key elements of CAT including reciprocal roles and reformulation to inform care planning and case management. The proposed study expands on the existing evidence base by utilising a comparator; a treatment as usual condition. The proposed mixed methods feasibility study will compare outcomes for both patients and care coordinators to assess the effectiveness of the intervention compared to controls in a community mental health team.

ELIGIBILITY:
Inclusion Criteria:

1. they are indicated as unsuitable for individual therapy,
2. there is a poor or challenging relationship between the patient and the care coordinator(s)
3. the care coordinator(s) feels a sense of 'stuckness' with the case
4. the patient is chaotic

Exclusion Criteria:

1. actively psychotic
2. severely misusing substances
3. have poor appointment attendance
4. indicating that they are actively suicidal and unwilling to commit to trying to stay safe.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Personality Structure Questionnaire (PSQ) | Screening (point of referral), start of waiting list (up to 2 weeks), end of waiting list (up to 12 weeks), start of treatment (up to 12 weeks), end of treatment (up to 22 weeks), 8 week follow-up (up to 30 weeks), 12 week follow-up (up to 34 weeks)
  Primary outcome measure for patients utilised to measure change across multiple time-points.
  The PSQ is an 8-item measure of identity disturbance. Each item is rated using a 5-point Likert scale. The maximum score on the scale is 40, indicating a high level of identity disturbance.
Perceived competence scale | Screening (point of referral), start of waiting list (up to 2 weeks), end of waiting list (up to 12 weeks), start of treatment (up to 12 weeks), end of treatment (up to 22 weeks), 8 week follow-up (up to 30 weeks), 12 week follow-up (up to 34 weeks)
  Primary outcome measure for care coordinators utilised to measure change across multiple time-points.
  The Perceived Competence Scale is a four item Likert-scale ranging from 1 to 7. The maximum score for each item is 7, and the maximum overall score for the scale is 28, indicating the highest levels of perceived competence.

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation (CORE-10) | Screening (point of referral), start of waiting list (up to 2 weeks), end of waiting list (up to 12 weeks), start of treatment (up to 12 weeks), end of treatment (up to 22 weeks), 8 week follow-up (up to 30 weeks), 12 week follow-up (up to 34 weeks)
  Secondary outcome measure for patients utilised to measure change across multiple time-points.
  The CORE-10 is a ten item questionnaire which measures psychological distress. The maximum score on this measure is 40, indicating the highest level of psychological distress.
Working Alliance Inventory Short-Revised (WAI-SR) | Screening (point of referral), start of waiting list (up to 2 weeks), end of waiting list (up to 12 weeks), start of treatment (up to 12 weeks), end of treatment (up to 22 weeks), 8 week follow-up (up to 30 weeks), 12 week follow-up (up to 34 weeks)
  Secondary outcome measure for patients utilised to measure change across multiple time-points.
  The WAI-SR is a 12 item scale; items are rated using a 5-point Likert scale. The items can be divided into three constructs, measuring goals, tasks and bond. Each of these domains have scores ranging from 5 to 20. Higher scores indicate better working alliance.
Doubt Subscale of the Mental Health Professionals Stress Scale (MHPSS) | Screening (point of referral), start of waiting list (up to 2 weeks), end of waiting list (up to 12 weeks), start of treatment (up to 12 weeks), end of treatment (up to 22 weeks), 8 week follow-up (up to 30 weeks), 12 week follow-up (up to 34 weeks)
  Secondary outcome measure for care coordinators utilised to measure change across multiple time-points.
  The doubt subscale is a six-item scale which measures professionals' doubt about their practice. Each item will be scored as 1 if present with a maximum score of 6, indicating high levels of doubt.

CONTACTS AND LOCATIONS:
Locations (1):
- Rotherham Doncaster and South Humber NHS Foundation Trust, Rotherham, United Kingdom

IPD SHARING:
Plan to Share IPD: No